CLINICAL TRIAL: NCT02284165
Title: Comparative Effectiveness of Rehabilitation Services for Survivors of Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00044034
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: retrospective analysis — Analysis of data for patients hospitalized in 2006-2008 with acute ischemic stroke, and successfully linked with Medicare claims through 2009

SUMMARY:
Retrospective analysis of Get With the Guidelines-Stroke data linked with Medicare claims and the AVAIL longitudinal data sets to assess patterns, predictors, and outcomes associated with the use of rehabilitation services following hospitalization for ischemic stroke. Primary completion defined as the end of primary analyses, consistent with the end of the PCORI Cycle I grant period. Study completion defined as acceptance of final research report and lay abstract by PCORI.

DETAILED DESCRIPTION:
The investigators will seek to answer three questions:

1. What are the person- and system-level factors associated with use of rehabilitation services following acute ischemic stroke?
2. Among stroke survivors discharged to short-term inpatient rehabilitation, are high-intensity services performed at an Inpatient Rehabilitation Facility (IRF) more effective than lower intensity services performed at a Skilled Nursing Facility (SNF), at improving patient outcomes at 3 and 12 months?
3. Among stroke survivors discharged home, is early follow-up with a physician more effective than follow-up after 7 days at 3 and 12 months?

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke within the Get With the Guidelines-Stroke data set for 2006-2008, and successfully linked to Medicare claims through 2009

Exclusion Criteria:

* death during index hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized for acute ischemic stroke in 2006-2008, and successfully linked to Medicare claims available through 2009
Sampling Method: Non-Probability Sample
Enrollment: 164246 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Bettger, ScD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xian Y, Thomas L, Liang L, Federspiel JJ, Webb LE, Bushnell CD, Duncan PW, Schwamm LH, Stein J, Fonarow GC, Hoenig H, Montalvo C, George MG, Lutz BJ, Peterson ED, Bettger JP. Unexplained Variation for Hospitals' Use of Inpatient Rehabilitation and Skilled Nursing Facilities After an Acute Ischemic Stroke. Stroke. 2017 Oct;48(10):2836-2842. doi: 10.1161/STROKEAHA.117.016904. Epub 2017 Aug 22. PMID 28830975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Starting population = 164,246 acute ischemic stroke patients with data in Get With the Guidelines linked to Medicare fee-for-service (FFS) claims. This was a retrospective analysis of existing data, so there were no patient milestones.
Pre-assignment Details: The following exclusions were applied prior to group assignment: death during index admission (n=10,466); loss of FFS eligibility not due to death during follow-up (n=1683); discharged to Federal hospital (n=102); transferred to another acute care hospital or discharged directly to nursing home for long-term care (n=4279).
Groups:
- Inpatient Rehab Facility (IRF): Discharged from hospital to inpatient rehabilitation facility
- Skilled Nursing Facility (SNF): Discharged from hospital to skilled nursing facility
- Discharged Home: Discharged from hospital to home with or without services
Period: Overall Study
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF) | Discharged Home
Started | 36448 | 40272 | 70996
Completed | 36448 | 40272 | 70996
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Acute ischemic stroke patients in the Get With the Guidelines registry with Medicare fee-for-service health insurance. Differentiation into study arms by discharge location meets the first primary aim of the study, to describe rehab service use through 90 days.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF) | Discharged Home | Total
Number analyzed (Participants) | 36448 | 40272 | 70996 | 147716
Age, Continuous [Median (Inter-Quartile Range); unit: years] — All analyses calculated by comparing only non-missing values.
  years | 79 [73 to 84] | 83 [73 to 88] | 78 [71 to 84] | 80 [74 to 86]
Sex/Gender, Customized [Number; unit: participants] — All analyses calculated by comparing only non-missing values. Gender missing among 5 patients discharged to IRF, and 2 patients discharged to SNF.
  participants
    Female | 20570 | 26801 | 38726 | 86097
    Male | 15873 | 13469 | 32270 | 61612
    Missing | 5 | 2 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All analyses calculated by comparing only non-missing values.
  Participants
    Hispanic or Latino | 1358 | 1231 | 2576 | 5165
    Not Hispanic or Latino | 35090 | 39041 | 68420 | 142551
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — All analyses calculated by comparing only non-missing values. Hispanic ethnicity collected as a category under Race, prior to revision of collection standards to match NIH/OMB.
  participants
    American Indian or Alaska Native | 74 | 43 | 110 | 227
    Asian | 508 | 580 | 1091 | 2179
    Native Hawaiian or Other Pacific Islander | 67 | 56 | 135 | 258
    Black or African American | 1358 | 1231 | 2576 | 5165
    White | 29720 | 33087 | 58290 | 121097
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 4721 | 5275 | 8794 | 18790
Region of Enrollment [Number; unit: participants]
  United States | 36448 | 40272 | 70996 | 147716

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Inpatient, Home, or Community Based Rehabilitation Services
Description: Received either inpatient care in an inpatient rehabilitation or skilled nursing facility, or home or community-based rehabilitation.
Time Frame: discharge through 90 days
Population: Acute ischemic stroke patients in the Get With the Guidelines registry with Medicare fee-for-service health insurance, analyzed as one cohort rather than by arm to differentiate the different types of rehabilitation services within the full patient population.
Measure: Number; unit: participants
Groups:
- All Patients: Examined descriptively for all patients in the study in order to differentiate the different types of rehabilitation services for the full stroke patient population.
Arm/Group | All Patients
Number analyzed (Participants) | 162432
participants
  Short-term inpatient rehab (inpt, skilled nurs.) | 76720
  Home or community-based rehab | 32350

2. Primary Outcome: Home-time
Description: Number of days alive and living outside of inpatient care
Time Frame: 12 months post-discharge
Population: Acute ischemic stroke patients in the Get With the Guidelines registry with Medicare fee-for-service health insurance, discharged to inpatient rehab or skilled nursing care and without survival limitations identified in-hospital. 69,212 patients met these criteria.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF)
Number analyzed (Participants) | 34815 | 34397
days | 271.2 (112.5) | 195.5 (138.5)

3. Secondary Outcome: Number of Participants Who Were Functionally Dependent or Dead 12 Months After Hospital Discharge
Description: 12-month functional status as measured by modified Rankin scale scores ranging between 0 (no symptoms) and 6 (death), among patients discharged to inpatient rehabilitation or skilled nursing facility. Outcome measure reports number of participants with Rankin score of 3-6. The outcome was not assessed among patients discharged home.
Time Frame: 12 months post-discharge
Population: Acute ischemic stroke patients in the Get With the Guidelines registry discharged to inpatient rehabilitation or skilled nursing facility, without survival limitations identified in-hospital and with 12-month follow-up as part of the Adherence Evaluation After Ischemic Stroke Longitudinal (AVAIL) registry. 473 participants met these criteria.
Measure: Number; unit: participants
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF)
Number analyzed (Participants) | 345 | 128
participants | 203 | 77

4. Secondary Outcome: Quality of Life (QOL)
Description: EuroQOL-5 Dimensions (EQ-5D) to assess health-related quality of life by asking and scoring the level of severity (1 = no problems, 2 = some problems, 3 = extreme problems) in 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Score for each question is added together to provide total score, which is converted to provide a range from 1 (maximum and highest health state for quality of life) down to 0 (lowest health state and quality of life).
Time Frame: 12 months post-discharge
Population: Acute ischemic stroke patients in the Get With the Guidelines registry discharged to inpatient rehabilitation or skilled nursing facility, without survival limitations identified in-hospital and with 12-month follow-up as part of the Adherence Evaluation After Ischemic Stroke Longitudinal (AVAIL) registry. 323 patients met these criteria.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF)
Number analyzed (Participants) | 239 | 84
units on a scale | 0.76 [0.46 to 0.84] | 0.68 [0.00 to 0.83]

5. Secondary Outcome: Number of Participants Who Were Institutionalized in a Nursing Home for Long-term Care Within 12 Months of Hospital Discharge.
Description: Institutionalization (primary living location in a nursing home for long-term care and not for rehabilitation or short-term skilled stay) as measured by patient or proxy family member report on 12-month follow-up phone call.
Time Frame: 12 months post-discharge
Population: Acute ischemic stroke patients in the Get With the Guidelines registry discharged to inpatient rehabilitation or skilled nursing facility, without survival limitations identified in-hospital and with 12-month follow-up as part of the Adherence Evaluation After Ischemic Stroke Longitudinal (AVAIL) registry. 473 patients met these criteria.
Measure: Number; unit: participants
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF)
Number analyzed (Participants) | 345 | 128
participants | 64 | 60

6. Secondary Outcome: Number of Participants Who Were Rehospitalized or Died Within 12 Months of Stroke Hospitalization.
Description: All-cause rehospitalization or death within 12 months of index stroke hospitalization as indicated in Medicare claims files.
Time Frame: 12 months post-discharge
Population: Acute ischemic stroke patients in the Get With the Guidelines registry with Medicare fee-for-service health insurance, discharged to inpatient rehabilitation or skilled nursing facility and without survival limitations identified in-hospital. 69,212 patients met these criteria.
Measure: Number; unit: participants
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF)
Number analyzed (Participants) | 34815 | 34397
participants | 18884 | 23411

7. Secondary Outcome: Number of Participants Who Died Within 12 Months of Stroke Hospitalization
Description: Death within 12 months of discharge from index stroke hospitalization as indicated in Medicare claims files
Time Frame: 12 months post-discharge
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Inpatient Rehab Facility (IRF) | Skilled Nursing Facility (SNF)
Number analyzed (Participants) | 34815 | 34397
participants | 6221 | 13274

ADVERSE EVENTS:
Description: This was a retrospective analysis of pre-existing data for acute ischemic stroke patients in the Get With the Guidelines registry with Medicare fee-for-service health insurance, or with 12-month follow-up as part of the Adherence Evaluation After Ischemic Stroke Longitudinal (AVAIL) registry. Adverse events were not assessed.
Groups:
- All Patients: Not applicable. This was a retrospective analysis of pre-existing data for acute ischemic stroke patients in the Get With the Guidelines registry with 12-month follow-up as part of the Adherence Evaluation After Ischemic Stroke Longitudinal (AVAIL) registry.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No